CLINICAL TRIAL: NCT00091312
Title: Randomized Phase III Intergroup Trial in Resected Stage 2 (Dukes B) Colon Cancer: 6-Month Infusional 5FU-CPT11 (+/- Folinic Acid) Versus Observation - Determination of Biologic Predictive and Response Factors
Brief Title: Fluorouracil and Irinotecan With or Without Leucovorin Compared With Observation in Treating Patients Who Have Undergone Surgery for Stage II Colon Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Federation Francophone de Cancerologie Digestive (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000387797; FFCD-EORTC-40012; EORTC-40012; PETACC-4
Record Dates: First submitted 2004-09-07; First posted 2004-09-09 (Estimated); Last update posted 2009-02-09 (Estimated); Status verified 2006-12

CONDITIONS: Colorectal Cancer
Keywords: stage II colon cancer; adenocarcinoma of the colon
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms | interventions — Fluorouracil; Irinotecan; Leucovorin; Chemotherapy, Adjuvant

INTERVENTIONS:
Drug: FOLFIRI regimen
Drug: fluorouracil
Drug: irinotecan hydrochloride
Drug: leucovorin calcium
Procedure: adjuvant therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as irinotecan, leucovorin, and fluorouracil, work in different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug and giving them after surgery may kill any remaining tumor cells. It is not yet known whether combination chemotherapy is more effective than observation alone in treating patients who have undergone surgery for colon cancer.

PURPOSE: This randomized phase III trial is studying irinotecan and fluorouracil with or without leucovorin to see how well they work compared to observation alone in treating patients who have undergone surgery for stage II colon cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare 5-year disease-free survival in patients with resected stage II adenocarcinoma of the colon treated with adjuvant chemotherapy comprising fluorouracil and irinotecan with or without leucovorin calcium vs no adjuvant therapy.

Secondary

* Compare 8-year overall survival in patients treated with these regimens.
* Compare tolerability of these regimens in these patients.
* Correlate clinical, histological, and biological prognostic factors with outcome in patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to participating center, disease stage (pT3 vs pT4), pathological differentiation (poorly or undifferentiated vs well or moderately differentiated), and microsatellite instability (positive vs negative vs unknown). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients are further randomized to receive 1 of 3 adjuvant chemotherapy regimens.

  * Regimen A: Patients receive irinotecan IV over 90 minutes followed by leucovorin calcium IV over 2 hours and fluorouracil IV continuously over 46 hours on days 1, 15, and 29. Treatment repeats every 42 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.
  * Regimen B: Patients receive irinotecan IV over 30-90 minutes followed by leucovorin calcium IV over 2 hours and fluorouracil IV continuously over 24 hours on days 1, 8, 15, 22, 29, and 36. Treatment repeats every 56 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.
  * Regimen C: Patients receive irinotecan IV over 60 minutes followed by fluorouracil IV continuously over 48 hours on days 1, 8, 15, 22, 29, and 36. Treatment repeats every 42 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients undergo observation only. Patients are followed every 6 months.

PROJECTED ACCRUAL: A total of 1,976 patients (988 per treatment arm [247 each in regimens A and B of arm I and 494 in regimen C of arm I]) will be accrued for this study within 4.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the colon

  * Stage II disease (pT3, N0 or pT4, N0)

    * Penetration of the subserosa or serosa
    * No lymph node metastases

      * At least 12 lymph nodes analyzed
* More than 1 synchronous primary colon tumor allowed

  * Staging determined for the more advanced tumor
* Curative radical resection within the past 2-8 weeks required

  * Proximal, distal, and radical margins must be free of tumor (R0 resection)
* No rectal tumors

  * Gross distal margin of the primary tumor must lie above the peritoneal reflection
* No known familial adenomatous polyposis
* No hereditary nonpolyposis colorectal cancer
* No distant metastases

PATIENT CHARACTERISTICS:

Age

* 18 to 75

Performance status

* WHO 0-1

Life expectancy

* Not specified

Hematopoietic

* Granulocyte count ≥ 2,000/mm^3
* Platelet count ≥ 100,000mm^3
* Hemoglobin ≥ 10 g/dL

Hepatic

* Bilirubin < 1.25 times upper limit of normal (ULN)
* No known Gilbert's syndrome

Renal

* Creatinine < 1.25 times ULN

Cardiovascular

* No severe or uncontrolled coronary disease
* No severe heart failure
* No uncontrolled arterial hypertension
* No myocardial infarction within the past year
* No cerebral vascular accident within the past year
* Cardiac arrhythmia allowed provided patient is on proper anticoagulation therapy* NOTE: *Aspirin is not considered proper anticoagulation

Gastrointestinal

* No Gardner's syndrome
* No Turcot's syndrome
* No Crohn's disease
* No ulcerative colitis

Other

* No other prior malignancy except adequately treated basal cell skin cancer or carcinoma in situ of the cervix
* No other serious disease
* No contraindication to any study drugs
* No known allergy to leucovorin calcium
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for up to 6 months after study treatment

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* No prior radiotherapy

Surgery

* See Disease Characteristics

Other

* No other concurrent anticancer therapy
* No concurrent vitamin supplements containing folic acid

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1976 (Estimated)
Dates: Start 2004-06

PRIMARY OUTCOMES:
Disease-free survival at 5 years

SECONDARY OUTCOMES:
Overall survival at 8 years
Tolerability
Correlation of clinical, histological, and biological prognostic factors with outcome

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Bedenne, MD, Study Chair — Hopital Du Bocage
Locations (9):
- National Cancer Institute - Cairo, Cairo, Egypt
- France (2):
  - Centre Hospitalier Universitaire Ambroise Pare - Boulogne, Boulogne-Billancourt
  - Hopital Du Bocage, Dijon
- Medizinische Klinik I, Dresden, Germany
- Italy (3):
  - Ospedali Riuniti di Bergamo, Bergamo
  - Azienda Ospedaliero Careggi, Florence
  - Universita Degli Studi di Florence - Policlinico di Careggi, Florence
- Instituto Portugues de Oncologia Centro do Porto, S. A., Porto, Portugal
- Hospital Universitario de Elche, Elche Alicante, Spain